CLINICAL TRIAL: NCT04679064
Title: Randomized Phase III Trial on NIraparib-TSR-042 (Dostarlimab) vs Physician's Choice CHEmotherapy in Recurrent, Ovarian, Fallopian Tube or Primary Peritoneal Cancer Patients Not Candidate for Platinum Retreatment: NItCHE Trial (MITO 33)
Brief Title: Trial on NIraparib-TSR-042 (Dostarlimab) vs Physician's Choice CHEmotherapy in Recurrent, Ovarian, Fallopian Tube or Primary Peritoneal Cancer Patients Not Candidate for Platinum Retreatment
Acronym: NItCHE-MITO33
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3392
Record Dates: First submitted 2020-10-05; First posted 2020-12-22 (Actual); Last update posted 2021-08-27 (Actual); Status verified 2020-09

CONDITIONS: Ovarian Cancer
MeSH Terms: conditions — Ovarian Neoplasms | interventions — niraparib; dostarlimab; liposomal doxorubicin; Paclitaxel; Gemcitabine; Topotecan; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Phisician's choice of standard chemotherapy (Active Comparator): Chemotherapy at physician's choice between Pegylated Liposomal Doxorubicin 40 mg/mq iv q 28 Weekly Paclitaxel 80 mg/mq d 1,8,15 q 28 Gemcitabine 1000 mg/mq d 1,8,15 q 28 Topotecan 1.25 mg/mq day 1-5 q 21
  +/- Bevacizumab at defined scehedule
  Interventions: Drug: Pegylated liposomal doxorubicin; Drug: Paclitaxel; Drug: Gemcitabine; Drug: Topotecan; Drug: Bevacizumab
- Niraparib+Dostarlimab (Experimental): Dostarlimab 500 mg q 3W for the fist 4 cycles, 1000 mg q 6W thereafter + Niraparib 300 mg or 200 mg if platelet count <150,000 /μL and/or body weight <77kg QD po q 28
  Interventions: Drug: Niraparib; Drug: Dostarlimab

INTERVENTIONS:
Drug: Niraparib — PARP-inihibitor
  Other Names: Zejula
  Arms: Niraparib+Dostarlimab
Drug: Dostarlimab — PD-1 inihibitor
  Other Names: TSR-042
  Arms: Niraparib+Dostarlimab
Drug: Pegylated liposomal doxorubicin — Chemotherapy drug
  Arms: Phisician's choice of standard chemotherapy
Drug: Paclitaxel — Chemotherapy drug
  Arms: Phisician's choice of standard chemotherapy
Drug: Gemcitabine — Chemotherapy drug
  Arms: Phisician's choice of standard chemotherapy
Drug: Topotecan — Chemotherapy drug
  Arms: Phisician's choice of standard chemotherapy
Drug: Bevacizumab — Chemotherapy drug
  Other Names: Avastin
  Arms: Phisician's choice of standard chemotherapy

SUMMARY:
Randomized phase 3 trial evaluating niraparib plus dostarlimab vs chemotherapy at physician's choice in the treatment of recurrent ovarian, fallopian tube or primary peritoneal cancer patients for which platinum is not an option

DETAILED DESCRIPTION:
Randomized phase 3 trial evaluating niraparib plus dostarlimab vs chemotherapy at physician's choice in the treatment of recurrent ovarian, fallopian tube or primary peritoneal cancer patients for which platinum is not an option.

The patients must have received no more than 2 previous chemotherapy lines. Stratification factors will include HRD status, previous treatment with parp and anti PD-1/PDL-1 inhibitors, Bevacizumab treatment and PDL1 expression.

Patients will continue to receive niraparib until disease progression (determined using RECIST v.1.1 criteria and clinical criteria), unacceptable toxicity, death, withdrawal of consent, or lost to follow-up, whichever comes first. Patients will continue to receive dostarlimab for a maximum of 2 years, or until disease progression (determined using RECIST v1.1 criteria and clinical criteria), unacceptable toxicity, death, withdrawal of consent, lost to follow-up, whichever may come first. Dose interruption and/or reduction may be implemented at any time for any grade toxicity considered intolerable by the patient.

ELIGIBILITY:
Inclusion Criteria:

1. Participant must have recurrent ovarian, Fallopian tube or primary peritoneal cancer not candidate for platinum retreatment; and in particular

   * platinum resistant patients (platinum-free interval 1-6 months from last dose of platinum)
   * patients for which platinum is contraindicated because of previous allergic reactions or residual toxicity (i.e nephrotoxicity or neurotoxicity)
   * patients not able( in physician's opinion) to receive further platinum or not willing (in patients' opinion) to receive further platinum
2. Participant must have an Eastern Cooperative Oncology Group (ECOG) performance status of ≤ 1
3. Participants must have measurable disease or evaluable based on RECIST 1.1 (patients with only CA 125 increase without evidence of disease are not included).
4. Participant must be ≥ 18 years of age
5. Participant must have adequate organ function
6. Participant receiving corticosteroids may continue as long as their dose is stable for least 4 weeks prior to initiating protocol therapy.
7. Participant must agree to not donate blood during the study or for 90 days after the last dose of study treatment.
8. Participants must agree to provide tissue from a newly obtained core or excisional biopsy of a tumor lesion. Newly-obtained is defined as a specimen obtained up to 6 weeks (42 days) prior to initiation of treatment on Day 1.

   Subjects for whom newly-obtained samples cannot be provided (e.g. inaccessible or subject safety concern) may submit an archived specimen.
9. Female participant has a negative urine or serum pregnancy test within 7 days prior to taking study treatment if of childbearing potential and agrees to abstain from activities that could result in pregnancy from screening through 180 days after the last dose of study treatment, or is of nonchildbearing potential.
10. Participant must agree to not breastfeed during the study or for 180 days after the last dose of study treatment.
11. Participant must be able to understand the study procedures and agree to participate in the study by providing written informed consent

Exclusion Criteria:

1. Participant must not be simultaneously enrolled in any interventional clinical trial
2. Participants have received >2 previous CHT lines (previous treatment with parp inhibitors and/or anti check point inhibitors is allowed providing that at least 6 months from last treatment are intercurred)
3. Participant must not have had major surgery ≤ 3 weeks prior to initiating protocol therapy and participant must have recovered from any surgical effects.
4. Participant must not have received investigational therapy ≤ 4 weeks, or within a time interval less than at least 5 half-lives of the investigational agent, whichever is shorter, prior initiating protocol therapy.
5. Participant has had radiation therapy encompassing >20% of the bone marrow within 2 weeks; or any radiation therapy within 1 week prior to Day 1 of protocol therapy.
6. Participant must not have a known hypersensitivity to niraparib and dostarlimab components or excipients.
7. Participant must not have received a transfusion (platelets or red blood cells) ≤ 4 weeks prior to initiating protocol therapy.
8. Participant must not have received colony-stimulating factors (eg, granulocyte colony-stimulating factor, granulocyte macrophage colony-stimulating factor, or recombinant erythropoietin) within 4 weeks prior initiating protocol therapy.
9. Participant has had any known Grade 3 or 4 anemia, neutropenia or thrombocytopenia due to prior chemotherapy that persisted > 4 weeks and was related to the most recent treatment.
10. Participant must not have any known history of myelodysplastic syndrome (MDS) or acute myeloid leukemia (AML)
11. Participant must not have a serious, uncontrolled medical disorder, nonmalignant systemic disease, or active, uncontrolled infection. Examples include, but are not limited to, uncontrolled ventricular arrhythmia, recent (within 90 days) myocardial infarction, uncontrolled major seizure disorder, unstable spinal cord compression, superior vena cava syndrome, or any psychiatric disorder that prohibits obtaining informed consent
12. Participant must not have had diagnosis, detection, or treatment of another type of cancer ≤ 3 years prior to initiating protocol therapy (except basal or squamous cell carcinoma of the skin and cervical cancer that has been definitively treated)
13. Participant must not have known, symptomatic brain or leptomeningeal metastases
14. Patient experienced ≥ Grade 3 immune-related AE with prior immunotherapy, with the exception of non-clinically significant lab abnormalities.
15. Participant has a diagnosis of immunodeficiency or has received systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to initiating protocol therapy.
16. Participant has a known history of human immunodeficiency virus (type 1 or 2 antibodies).
17. Participant has known active hepatitis B (e.g., hepatitis B surface antigen [HBsAg] reactive) or hepatitis C (e.g., hepatitis C virus [HCV] ribonucleic acid [qualitative] is detected).
18. Participant has an active autoimmune disease that has required systemic treatment in the past 2 years (ie, with use of disease-modifying agents, corticosteroids, or immunosuppressive drugs). Replacement therapy (eg, thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
19. Participant must not have a history of interstitial lung disease.
20. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
21. Has received a live vaccine within 30 days of planned start of study therapy. Note: Seasonal influenza vaccines for injection are generally inactivated flu vaccines and are allowed; however intranasal influenza vaccines are live attenuated vaccines, and are not allowed.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 427 (Estimated)
Dates: Start 2020-12-01 (Actual); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
Overall Survival | 4 years
  The length of time from tfrom the date of randomization to the date of death by any cause

SECONDARY OUTCOMES:
Progression free survival | 4 years
  the length of time from the date of randomization to the earlier date of assessment of progression or death by any cause in the absence of progression.
Time to first subsequent therapy | 4 years
  The length of the time interval from the date of randomization to earliest date of fist subsequent therapy or death
Response rate | 4 years
  the percentage of patients with CR or PR, as assessed by RECIST (Response Evaluation Criteria on Solid Tumor) v.1.1 criteria evaluated by the investigator.
Number and type of adverse events | 4 years
  Safety and tolerability of patients receiving chemotherapy or dostarlimab plus niraparib evaluated according to CTCAE vers 5.0.
Patient-reported outcomes for physical well-being | 4 years
  quality of life of patients, in terms of physical well-being, evaluated using EORTC (European Organization for Research and Treatment of Cancer) QLQ C30 (Quality of life Questionnaires C30). "1" is the minimum score and is the better outcome, "4" is the maximum score and is the worse outcome.
Patient-reported outcomes for physical well-being | 4 years
  quality of life of patients, in terms of physical well-being, evaluated using EORTC (European Organization for Research and Treatment of Cancer) QLQ OV28 (Quality of life Questionnaires OV28). "1" is the minimum score and is the better outcome, "4" is the maximum score and is the worse outcome.
Patient-reported outcomes for physical well-being | 4 years
  quality of life of patients, in terms of physical well-being, evaluated using EQ-5DL (EURO-QOL). "0" is the minimum score and is the worse outcome, "100" is the maximum score and is the better outcome.
Patient-reported outcomes for social/family well-being | 4 years
  quality of life of patients, in terms of social/family well-being, evaluated using EORTC (European Organization for Research and Treatment of Cancer) QLQ C30 (Quality of life Questionnaires C30). "1" is the minimum score and is the better outcome, "4" is the maximum score and is the worse outcome.
Patient-reported outcomes for social/family well-being | 4 years
  quality of life of patients, in terms of social/family well-being, evaluated using EORTC (European Organization for Research and Treatment of Cancer) QLQ OV28 (Quality of life Questionnaires OV28). "1" is the minimum score and is the better outcome, "4" is the maximum score and is the worse outcome.
Patient-reported outcomes for social/family well-being | 4 years
  quality of life of patients, in terms of social/family well-being, evaluated using EORTC (European Organization for Research and Treatment of Cancer) EQ-5DL (EURO-QOL). "0" is the minimum score and is the worse outcome, "100" is the maximum score and is the better outcome.
Patient-reported outcomes for emotional well-being | 4 years
  quality of life of patients, in terms of emotional well-being, evaluated using EORTC (European Organization for Research and Treatment of Cancer) QLQ C30 (Quality of life Questionnaires C30). "1" is the minimum score and is the better outcome, "4" is the maximum score and is the worse outcome.
Patient-reported outcomes for emotional well-being | 4 years
  quality of life of patients, in terms of emotional well-being, evaluated using EORTC (European Organization for Research and Treatment of Cancer) QLQ OV28 (Quality of life Questionnaires OV28). "1" is the minimum score and is the better outcome, "4" is the maximum score and is the worse outcome.
Patient-reported outcomes for emotional well-being | 4 years
  quality of life of patients, in terms of emotional well-being, evaluated using EORTC (European Organization for Research and Treatment of Cancer) EQ-5DL (EURO-QOL). "0" is the minimum score and is the worse outcome, "100" is the maximum score and is the better outcome.

CONTACTS AND LOCATIONS:
Locations (8):
- Italy (8):
  - Azienda Ospedaliera Spedali Civili, Brescia
  - Istituto Tumori della Romagna IRST IRCCS, Meldola
  - IEO-Istituto Europeo di Oncologia, Milan
  - IRCCS Ospedale San Raffaele, Milan
  - Istituto Nazionale Tumori IRCCS Fondazione G. Pascale, Naples
  - Nuovo Ospedale degli Infermi, Ponderano
  - Fondazione Policlinico Universitario Agostino Gemelli IRCCS, Rome
  - Istituti fisioterapici Ospitalieri - Istituto Tumori Regina Elena, Rome

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Musacchio L, Salutari V, Pignata S, Braicu E, Cibula D, Colombo N, Frenel JS, Zagouri F, Carbone V, Ghizzoni V, Giolitto S, Giudice E, Perri MT, Ricci C, Scambia G, Lorusso D. Randomized phase III trial on niraparib-TSR-042 (dostarlimab) versus physician's choice chemotherapy in recurrent ovarian, fallopian tube, or primary peritoneal cancer patients not candidate for platinum retreatment: NItCHE trial (MITO 33). Int J Gynecol Cancer. 2021 Oct;31(10):1369-1373. doi: 10.1136/ijgc-2021-002593. PMID 34607820